CLINICAL TRIAL: NCT03617341
Title: Brain Monitoring for High Risk of Brain Metastases in Metastatic Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2018-0254
Record Dates: First submitted 2018-07-17; First posted 2018-08-06 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Metastatic Breast Cancer With HER2 Positive; Triple Negative Breast Cancer
Keywords: Breast cancer; brain metastases; screening; brain MRI
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Breast Neoplasms; Brain Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Brain MRI: Regular brain MRI can detect early brain metastases in metastatic Breast cancer with high risk subgroups, such as HER2-positive and triple negative.
  Interventions: Procedure: Brain MRI

INTERVENTIONS:
Procedure: Brain MRI — Brain MRI will be taken at the time of initial diagnosis, first- and second-line treatment failure. Therefore, the investigators expect that early detection of brain metastases before the onset of symptoms will affect the overall prognosis of MBC patients.

SUMMARY:
In general, brain metastases found after development of neurologic symptoms have poor prognosis. Therefore, the investigators aim to investigate whether regular brain MRI (Magnetic Resonance Imaging) can detect early brain metastases and influence survival through early brain management in HER2-positive and triple negative breast cancer.

DETAILED DESCRIPTION:
It is well known that HER2-receptor positive and triple negative metastatic breast cancer (MBC) have poor prognosis than hormone receptor positive metastatic breast cancer. However, as new therapies such as trastuzumab and pertuzumab are introduced, overall survival was extended in patients with metastatic breast cancer compared with the previous 10 years. As a result, the number of breast cancer patients with brain metastases has increased, the demand for treatments of brain metastases is increasing.

The incidence of brain metastases in MBC has been reported to be 7.6% and 10.8% in luminal A / B, respectively. However, HER2-positive and triple negative breast cancer with the incidence of more than 30% of brain metastases were at high risk group of brain metastases.

In general, brain metastases found after development of neurologic symptoms have poor prognosis. Therefore, the investigators aim to investigate whether regular brain MRI (Magnetic Resonance Imaging) can detect early brain metastases and influence survival through early brain management in HER2-positive and triple negative breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 19 years
* Pathologically documented breast cancer that:

  1. is unresectable or metastatic ;
  2. has confirmed HER2 positive expression according to American Society of Clinical Oncology- College of American Pathologists (ASCO-CAP) guidelines or triple negative breast cancer
* No prior systemic palliative treatment of metastatic breast cancer
* Must have provided informed consent for study participation before performance of any study-specific procedures or tests

Exclusion Criteria:

* History of prior treatments about brain metastases or leptomeningeal metastases
* Symptomatic brain metastases at screening period
* Has received more than second-line systemic treatments (including endocrine therapy)
* For subjects who have difficulty lying down or who have claustrophobia, they can undergo sedation during brain MRI
* History of hypersensitivity reaction to contrast or drug allergic reaction
* Patients who inserted metallic prosthesis (pacemaker, denture, hearing aid, aneurysm clip, metallic material of eyeball, artificial joint, insulin pump, chemo-port, temporary tissue expander for breast reconstruction, etc) can be conducted after consultation with investigator before MRI.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Social, familial, or geographical factors that would interfere with study participation or follow-up

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were initial diagnosed with HER2-positive, triple negative metastatic breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-10-02 (Actual); Primary Completion 2021-07-30 (Estimated); Study Completion 2023-06-03 (Estimated)

PRIMARY OUTCOMES:
The incidence rates of brain metastases with high risk patients in metastatic breast cancer | 5 years
  The incidence rates of brain metastases with high risk patients in metastatic breast cancer at initial diagnosis and failure of first- and second-line treatments confirmed by brain MRI

SECONDARY OUTCOMES:
The incidence rate of brain oligometastasis (≤ 4) confirmed by brain MRI | 5 years
  To evaluate the incidence rate of brain oligometastsais (≤ 4) confirmed by brain MRI
Intracranial progression free survival(PFS) after treatment of brain metastases | 5 years
  To evaluate intracranial progression free survival(PFS) after treatment of brain metastases
The overall survival (OS) after diagnosis to brain metastases | 5 years
  To evaluate the overall survival (OS) after diagnosis to brain metastases
The period from diagnosis to treatment of brain metastases | 5 years
  To evaluate the period from diagnosis to treatment of brain metastases
The cognitive impairment assessment after brain metastases | 5 years
  To evaluate the cognitive impairment assessment after brain metastases

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei Cancer Center, Severance Hospital, Yonsei University Health System, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided